CLINICAL TRIAL: NCT01547260
Title: Phase I/II Study of Lenalidomide and Gemcitabine as First-line Treatment in Patients With Locally Advanced or Metastatic Pancreatic Cancer
Brief Title: Lenalidomide and Gemcitabine as First-line Treatment in Patients With Pancreatic Cancer
Acronym: LENAGEM
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Maria Liljefors (Other)
Collaborators: Karolinska University Hospital (Other); Karolinska Institutet (Other); Celgene (Industry)
Responsible Party: Sponsor-Investigator, Maria Liljefors, MD, Senior consultant, Karolinska University Hospital
Organization: Karolinska University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LENAGEM-PANC
Record Dates: First submitted 2012-02-28; First posted 2012-03-07 (Estimated); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Pancreatic Carcinoma Metastatic; Pancreatic Ductal Adenocarcinoma
MeSH Terms: interventions — Gemcitabine; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lenalidomide (Experimental): Phase I; Lenalidomide capsules will be taken orally each day on days 1-21 of each 28-day cycle. 3 subjects will be enrolled into each dose cohort for 15, 20 and 25 mg/day. Gemcitabine, 1000 mg/m2 in 0.9% sodium chloride will be administered iv over 30 minutes, at days 1, 8, 15 of each 28-day cycle. Phase II: Every other consecutive included subject in phase II part will be treated with either single lenalidomide (days 1-21 of 28) or single gemcitabine (days 1, 8, 15 of 28) during Cycle 1. The first included patient in phase II part will start with single lenalidomide. From treatment cycle number 2 and beyond, all subjects in the phase II part of the study will be treated with lenalidomide in combination with gemcitabine.
  Interventions: Drug: Gemzar
- gemcitabine (Experimental): Gemcitabine, 1000 mg/m2 in 0.9% sodium chloride will be administered iv over 30 minutes, at days 1, 8, 15 of each 28-day cycle in both phase I and II. Phase I:Lenalidomide capsules will be taken orally each day on days 1-21 of each 28-day cycle. 3 subjects will be enrolled into each dose cohort for 15, 20 and 25 mg/day. Phase II: Every other consecutive included subject in phase II part will be treated with either single lenalidomide (days 1-21 of 28) or single gemcitabine (days 1, 8, 15 of 28) during Cycle 1. The first included patient in phase II part will start with single lenalidomide. From treatment cycle number 2 and beyond, all subjects in the phase II part of the study will be treated with lenalidomide in combination with gemcitabine.
  Interventions: Drug: Revlimid

INTERVENTIONS:
Drug: Gemzar — Gemcitabine (Gemzar®), 1000 mg/m2 in 0.9% sodium chloride will be administered as intravenous infusion over 30 minutes, weekly for 3 weeks then rest for 1 week (days 1, 8, 15 of each 28-day cycle).
  Other Names: Revlimid
  Arms: Lenalidomide
Drug: Revlimid — Lenalidomide capsules will be taken orally in the morning each day on days 1-21 of each 28-day cycle. Phase I; Three subjects will be enrolled into each dose cohort for 15, 20 and 25 mg/day, respectively. Phase II; Lenalidomide at dose determined in Phase I, will be administered orally once daily for 21 days followed by 7 days rest.
  Other Names: Gemzar
  Arms: gemcitabine

SUMMARY:
The purpose of this study is to ascertain whether treatment with lenalidomide or lenalidomide in combination with gemcitabine induces modulation of immune effector functions and to characterize the nature of immune functions.

DETAILED DESCRIPTION:
Pancreatic cancer is characterised by aggressive growth, treatment resistance and an extremely poor prognosis. In subjects with locally advanced or metastatic disease, the median survival is approximately 6 - 11 months and 2 - 6 months, respectively. The currently accepted treatment for this disease in EU is gemcitabine which supplanted treatment with 5-FU after it was shown that median survival duration was marginally improved (4.41 and 5.65 months respectively, p = 0,022). The reported median survival time for subjects treated with single-agent gemcitabine in randomized phase III studies ranged form 4.9 to 7.2 months. Despite these improvements in the treatment of pancreatic cancer, the prognosis remains very poor. Lenalidomide (Revlimid®) belongs to a proprietary class of compounds called immunomodulatory drugs (IMiDs). IMiDshave both immunomodulatory and anti-angiogenic properties which could confer antitumour and antimetastatic effects. Lenalidomide has been demonstrated to possess anti-angiogenic activity through inhibition of bFGF, VEGF and TNF-alpha induced endothelial cell migration, due at least in part to inhibition of Akt phosphorylation response to bFGF.In addition, lenalidomide has a variety of immunomodulatory effects. Gemcitabine (Gemzar®) is a synthetic pyrimidine nucleoside analogue that is used as standard treatment of advanced pancreatic cancer. Beside the cytotoxic activity of gemcitabine, accumulating evidence has indicated that the product promote specific anticancer immune responses that contribute to the therapeutic effects of conventional therapy.Down-regulation in survival rate of pancreatic cell lines has more recently been observed, when treated with lenalidomide and gemcitabine in sub-optimal concentrations.Those data supports a hypothesis of a potential hyper-additive affect of the treatments given in combination. Therefore lenalidomide and gemcitabine should be of major interest to explore for combination therapy.

This is a phase I/II open-label, multi-center study. It will consist of a phase I dose-finding part and a phase II part during which subjects will be treated at the MTD established during phase I. Lenalidomide will be administered by a stepwise dose-escalation schedule in the phase I part. Thus, the primary endpoint in the phase I part is to determine the MTD and safety of the regimen lenalidomide and gemcitabine as first-line treatment in subjects with advanced pancreatic cancer.In the phase II part, primary endpoint is to evaluate the immunomodulatory effects of lenalidomide in combination with gemcitabine in the same patient population.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed, unresectable, locally advanced, or metastatic adenocarcinoma of the pancreas.
* ECOG performance status of 0 or 1, see Appendix 1.
* Life expectancy > 12 weeks.
* Must understand and voluntarily sign an informed consent form.
* Age > 18 years at the time of signing informed consent form.
* Must be able to adhere to the study visit schedule and other protocol requirements.
* Female subjects of childbearing potential† must:

  * Understand that the study medication is expected to have a teratogenic risk
  * Agree to use, and be able to comply with, effective contraception without interruption, 4 weeks before starting study drug, throughout study drug therapy (including dose interruptions) and for 4 weeks after the end of study drug therapy, even if she has amenorrhoea
* Male subjects must:

  * Agree to use condoms throughout study drug therapy, during any dose interruption and for one week after cessation of study therapy if their partner is of childbearing potential and has no contraception.
  * Agree not to donate semen during study drug therapy and for one week after end of study drug therapy

Exclusion Criteria:

* Prior use of systemic chemotherapy for the treatment of adenocarcinoma of the pancreas (with the exception of gemcitabine, fluorouracil, or capecitabine in the adjuvant setting).
* Laboratory abnormalities:
* Prior history of malignancy within 5 years (except basal or squamous cell carcinoma or carcinoma in situ of the cervix or breast, localized prostate cancer with PSA < 1,0 mg/dL).
* Subjects with a history of or active DVT or PE that are not therapeutically managed on a stable dose of appropriate anticoagulant.
* Brain metastases (subjects that are asymptomatic and do not require steroid control may be enrolled at the discretion of the investigator).
* Surgery within 28 days prior to cycle 1 Day 1 (minimally invasive procedures for the purpose of diagnosis or staging of the disease are permitted, including stent placement and insertion of central venous access advice).
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
* Any serious medical condition or psychiatric illness that places the subject at an unacceptable risk for study participation or would prevent the subject from signing the informed consent form.
* Prior therapy with lenalidomide or thalidomide.
* Use of any other experimental drug or therapy within 28 days prior to Cycle 1 Day 1.
* Pregnant or lactating females.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2009-10; Primary Completion 2014-01 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Safety (phase I). | Within the first day after start of treatment until 30 days post the last dose of study drug.
  In the phase I part of the study, the primary outcome is to determine the MTD and safety of the regimen lenalidomide and gemcitabine in combination. Data from all subjects who receive any study drug will be included in the safety analyses, according to the NCI CTCAE v3.0.
Immunomodulatory effect (phase II). | Within the first day of treatment until 60 days after start of treatment.
  In the phase II part, the primary endpoint is to evaluate assessment of immunological reaction.The changes in immune responses at the end of cycle 1 (single lenalidomide or single gemcitabine) and cycle 2 (lenalidomide combined with gemcitabine) will be described in relation to baseline within the individual patient.

SECONDARY OUTCOMES:
Clinical efficacy | Within start of treatment until start of therapy until clinical and/or radiological signs of progression of the disease by treatment group together.
  Progression-free survival (PFS) will be presented as time from start of therapy until clinical and/or radiological signs of progression of the disease by treatment group together.
  Survival rate at 12 months will be presented as rate of patients still alive at 12 months after start of therapy by treatment group together.
  Overall survival (OS) will be presented as time from start of therapy until death by treatment group together.

CONTACTS AND LOCATIONS:
Overall Officials: Håkan Mellstedt, Prof., Principal Investigator — Karolinska University Hospital
Locations (1):
- Karolinska University Hospital, Stockholm, Solna, Sweden

REFERENCES:
- [Derived] Ullenhag GJ, Mozaffari F, Broberg M, Mellstedt H, Liljefors M. Clinical and Immune Effects of Lenalidomide in Combination with Gemcitabine in Patients with Advanced Pancreatic Cancer. PLoS One. 2017 Jan 18;12(1):e0169736. doi: 10.1371/journal.pone.0169736. eCollection 2017. PMID 28099502
- [Derived] Ullenhag GJ, Rossmann E, Liljefors M. A phase I dose-escalation study of lenalidomide in combination with gemcitabine in patients with advanced pancreatic cancer. PLoS One. 2015 Apr 2;10(4):e0121197. doi: 10.1371/journal.pone.0121197. eCollection 2015. PMID 25837499